CLINICAL TRIAL: NCT02140749
Title: Randomized, Placebo-controlled Double-blind Cross-over Study to Evaluate the Effects of Short-chain Fructooligosaccharides on Stool Frequency in Constipated Subjects
Brief Title: Trial on Short-chain Fructooligosaccharides, Microbiota, and Constipation in Adults
Acronym: TOMCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NL46640.081.14
Record Dates: First submitted 2014-04-24; First posted 2014-05-16 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Functional Constipation
Keywords: Bifidobacteria; Bristol Stool Scale; Constipation; Diet; Fructooligosacchardes; Microbiota; Oligofructose
MeSH Terms: conditions — Constipation | interventions — oligofructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- sc-FOS 2g/day (Experimental): Placebo (4 weeks) Short-chain fructooligosaccharide 2 g/day (4 weeks)
  Interventions: Dietary Supplement: sc-FOS 2g/day; Dietary Supplement: Placebo
- sc-FOS 4g/day (Experimental): Placebo (4 weeks) Short-chain fructooligosaccharide 4 g/day (4 weeks)
  Interventions: Dietary Supplement: sc-FOS 4g/day; Dietary Supplement: Placebo
- sc-FOS 8g/day (Experimental): Placebo (4 weeks) Short-chain fructooligosaccharide 8 g/day (4 weeks)
  Interventions: Dietary Supplement: sc-FOS 8g/day; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: sc-FOS 2g/day — Chewing tablets containing Short-chain fructooligosaccharides 2g/day
  Other Names: FOS; Oligofructose; scFOS; Short-chain fructo-oligosaccharide
  Arms: sc-FOS 2g/day
Dietary Supplement: sc-FOS 4g/day — Chewing tablets containing short-chain Fructooligosaccharides 4g/day
  Other Names: FOS; Oligofructose; scFOS; Short-chain fructo-oligosaccharide
  Arms: sc-FOS 4g/day
Dietary Supplement: sc-FOS 8g/day — Chewing tablets containing short-chain Fructooligosaccharides 8g/day
  Other Names: FOS; Oligofructose; scFOS; Short-chain fructo-oligosaccharide
  Arms: sc-FOS 8g/day
Dietary Supplement: Placebo — Chewing tablets without short-chain Fructooligosaccharides

SUMMARY:
Rationale: The dietary short-chain fructooligosaccharides have been shown to increase fecal bacterial mass and fermentation metabolites which might stimulate gut motility. Therefore, these dietary non-digestible carbohydrates might relieve functional constipation.

Objective: Study the effect of short-chain fructooligosaccharides on functional constipation.

Study design: A 16-week, randomized, placebo-controlled, double-blind cross-over trial with intervention periods of 4 weeks with a run-in period of 4 weeks and a wash-out period of 4 weeks.

Study population: Human subjects with functional constipation according to ROMEIII criteria (total n=120; male and female; 18-75 yr).

Intervention: Placebo and one out of 3 dosages of short-chain fructo-oligosaccharides, (Degree of Polymerisation of 3-5; 2, 4 and 8 g/day) for 4 weeks. scFOS will be given as oral chews.

Main study parameters: The primary parameter is the number of complete bowel movements per day in subjects with functional constipation according to Rome III criteria. Secondary outcomes are Stool consistency (Bristol Stool Scale), Stool frequency, Severity of symptoms (Constipation Scoring System; CSS) and Quality of Life (Patient Assessment of Constipation Quality of Life; PAC-QoL).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 yr
* Agree to study design (signed informed consent)
* At least two of the following symptoms ≥25% of the time with criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to inclusion (ROME III criteria for functional constipation):

  * straining, lumpy or hard stool
  * sensation of incomplete evacuation
  * sensation of anorectal obstruction ⁄ blockage
  * use of manual manoeuvres
  * <3 bowel movements per week
* Availability of internet connection
* BMI 20-30
* Male or female
* Willingness to abstain from functional ingredients and such as probiotics, prebiotics and foods containing high amounts of fermentable fibers and laxatives starting 1 month prior to start of the study as well as during the washout period.

Exclusion Criteria:

* Currently participating in another clinical trial
* Drug usage
* Excessive alcohol usage (>4 consumptions/day or >20 consumptions/week)
* Pregnancy or lactating
* Underlying disease of the GI-tract or previous laparotomy, except cholecystectomy and appendectomy
* Use of antibiotics within 1 month prior to inclusion
* Vegetarians
* Weight loss > 5 kg within 1 month prior to inclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stool frequency (Number of complete bowel movements per day) | Change over week 4 and week 12

SECONDARY OUTCOMES:
Stool consistency (Bristol Stool Scale) | Change over week 4 and week 12
Severity of symptoms (Constipation Scoring System; CSS) | Change over week 4 and week 12
Quality of Life (Patient Assessment of Constipation Quality of Life; PAC-QoL) | Change over week 4 and week 12

CONTACTS AND LOCATIONS:
Overall Officials: Sandra ten Bruggencate, PhD, Principal Investigator — NIZO Food Research
Locations (1):
- NIZO food research, Ede, Gelderland, Netherlands

REFERENCES:
- See also: Related Info — http://www.nizo.com